CLINICAL TRIAL: NCT03766438
Title: Stories for Change: Digital Storytelling for Diabetes Self-Management Among Hispanic Adults
Acronym: S4C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Hennepin Healthcare (Other); Mountain Park Health Center - Phoenix, AZ (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mark L Wieland, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 18-002998; R01DK113999-01A1 (NIH)
Record Dates: First submitted 2018-11-27; First posted 2018-12-06 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will view the 12-minute digital storytelling intervention that has been previously pilot-tested, in addition to usual clinical care.
  Interventions: Behavioral: Digital Storytelling Intervention
- Control (No Intervention): The comparison group will receive usual clinical care.

INTERVENTIONS:
Behavioral: Digital Storytelling Intervention — 12-minute digital storytelling intervention in Spanish, with four individuals explaining their personal Type 2 Diabetes stories.
  Arms: Intervention

SUMMARY:
Hispanic adults are twice as likely to have type 2 diabetes mellitus (T2D) and 1.5 times more likely to die from the disease than non-Hispanic whites. These disparities are mediated, in part, by less healthful levels of physical activity, dietary quality, medication adherence, and self-monitoring of blood glucose than non-Hispanic whites. Innovative approaches that arise from affected communities are needed to address these health disparities.

Community-based participatory research (CBPR) has been successful in targeting health issues among Hispanic and immigrant populations; CBPR is an effective approach for addressing health behaviors in a sociocultural context. In 2004, the research team developed a CBPR partnership between immigrant communities and academic institutions called Rochester Healthy Community Partnership (RHCP)

Storytelling or narrative-based interventions are designed to incorporate culture-centric health messaging to promote behavior change among vulnerable populations. Digital storytelling interventions are narrative-based videos elicited through a CBPR approach to surface the authentic voices of individuals overcoming obstacles toward engaging in health promoting behaviors to shape positive health behaviors of viewers through influences on attitudes and beliefs.

RHCP partners from Hispanic communities identified T2D as a priority area for intervention, and have co-created each of the formative phases leading up to this proposal. Narrative theory and social cognitive theory formed the conceptual basis for intervention development. The study team conducted surveys and focus groups to derive the approach and personnel for building an authentic intervention that was created in a digital storytelling workshop where stories about diabetes self-management were captured, recorded, and edited to derive the final intervention products in video forma. The respective digital storytelling videos were pilot tested with 25 patients across healthcare institutions in Minnesota and Arizona. The intervention was rated as highly acceptable, culturally relevant, and perceived as efficacious for motivating behavioral change.

The overall objective of this project is therefore to assess the efficacy of a digital storytelling intervention derived through a CBPR approach on self-management of T2D among Hispanic adults.

DETAILED DESCRIPTION:
The study team will conduct a two-group randomized controlled trial in primary care clinical settings at two healthcare institutions among 450 Hispanic adults with poorly controlled T2D (hemoglobin A1c≥8%). The intervention group will view the 12-minute digital storytelling video. Both the intervention and comparison groups will receive diabetes education and resource cards, as well as usual clinical care. The primary outcome will be glycemic control as measured by hemoglobin A1c 3 months after intervention delivery. Secondary outcomes will include diabetes self-management behaviors, blood pressure, LDL-cholesterol, and body mass index. The impact of concomitant covariates, including sex, age, and socio-economic status, on the sensitivity of the intervention effect will also be explored.

ELIGIBILITY:
1. Self-identifies as Hispanic or Latino.
2. Between 18 and 70 years of age.
3. Receives primary care at the clinical site.
4. Visited the primary care site at least once in the least twelve months.
5. Intention to continue receiving care at the clinic for the next six months.
6. Diagnosis of T2D in medical record.
7. T2D diagnosis for six months or longer.
8. Most recent hemoglobin A1c≥8%.

Not eligible if someone in the same household is participating in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Wieland, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mountain Park Health Center, Phoenix, Arizona
  - Hennepin Healthcare, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Wieland ML, Vickery KD, Hernandez V, Ford BR, Gonzalez C, Kavistan S, Iteghete S, Patten CA, Njeru JW, Lohr AM, O'Byrne J, Novotny PJ, Singh DP, Larkey LK, Goodson M, Capetillo GP, Sia IG. Digital Storytelling Intervention for Hemoglobin A1c Control Among Hispanic Adults With Type 2 Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2424781. doi: 10.1001/jamanetworkopen.2024.24781. PMID 39093566
- [Derived] Lohr AM, Vickery KD, Hernandez V, Ford BR, Gonzalez C, Kavistan S, Patten CA, Njeru JW, Novotny PJ, Larkey LK, Singh D, Wieland ML, Sia IG. Stories for change protocol: A randomized controlled trial of a digital storytelling intervention for Hispanic/Latino individuals with type 2 diabetes. Contemp Clin Trials. 2023 Mar;126:107093. doi: 10.1016/j.cct.2023.107093. Epub 2023 Jan 20. PMID 36682492

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 227 | 224
Completed | 191 | 199
Not Completed | 36 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 227 | 224 | 451
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (9.25) | 54.5 (9.08) | 54.4 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 156 | 314
  Male | 69 | 68 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 227 | 224 | 451
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 227 | 224 | 451
Hemoglobin A1C [Mean (Standard Deviation); unit: Percent] | 9.1 (1.72) | 9.4 (1.75) | 9.25 (1.73)

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control as Measured by Hemoglobin A1c at Baseline and 3 Months
Description: The rationale for use of hemoglobin A1c as an indicator of diabetes control is based on national and regional data that demonstrate significant disparities in reaching hemoglobin A1c targets for Hispanic populations compared with non-Hispanic whites. The importance of glycemic control as part of the comprehensive management of diabetes is well documented, and hemoglobin A1c testing is a well-established strategy to monitor glycemic control in patients with diabetes.
Time Frame: Baseline and 3 months.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Intervention | Control
Number analyzed (Participants) | 191 | 199
Percent
  Baseline | 9.1 (1.7) | 9.4 (1.8)
  3 months | 8.4 (1.6) | 8.8 (2)

ADVERSE EVENTS:
Time Frame: Through study completion (6 months)
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/227 | 0/224
Serious Adverse Events (participants affected / at risk) | 0/227 | 0/224
Other Adverse Events (participants affected / at risk) | 0/227 | 0/224

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT03766438/Prot_SAP_000.pdf